CLINICAL TRIAL: NCT07189117
Title: Cancer and Immune Cell Metabolism in Patients With Hematological Malignancies
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01775;th25Aposotolova
Record Dates: First submitted 2025-09-05; First posted 2025-09-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy
Keywords: allo-HSCT
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood and Bone Marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with hematological cancers
- Healthy stem cell donors

SUMMARY:
This study investigates how metabolism in cancer and immune cells shapes the bone marrow environment, influences therapy resistance, and affects outcomes in hematological malignancies.

DETAILED DESCRIPTION:
Hematological malignancies, such as acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), and myelofibrosis, are aggressive cancers of the blood and immune system. While chemotherapy is commonly used, allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains the only curative option for many patients. Allo-HSCT relies on donor immune cells, particularly T cells, to eliminate residual malignant cells, but relapse occurs in a significant proportion of patients, underscoring the need for improved therapeutic strategies.

Recent research has highlighted the critical role of cellular metabolism in both cancer cell survival and immune cell function. AML cells, for example, rely on mitochondrial respiration, while immune cells are sensitive to metabolic changes in the bone marrow microenvironment. These metabolic interactions may influence disease progression, therapy resistance, and immune-mediated anti-tumor responses, yet they remain poorly understood.

The primary goal of this study is to investigate how cancer and immune cell metabolism shapes the bone marrow environment and influences treatment outcomes in patients with hematological malignancies. By performing detailed metabolic profiling of malignant cells, immune cells, and extracellular metabolites across disease stages and treatment time points, the study aims to identify key metabolic pathways and interactions that could serve as targets for novel therapies and guide personalized treatment approaches.

This research is expected to deepen the understanding of metabolic mechanisms underlying hematological cancers and allo-HSCT outcomes, potentially leading to improved strategies to enhance anti-tumor immunity, prevent relapse, and optimize patient-specific therapy.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* signed written informed consent
* For participants with hematological cancers: diagnosis of MDS, AML, ALL, PMF or post-ET/PV MF

Exclusion Criteria:

* pregnant or lactating women,
* inability to give consent,
* active malignant disease (other than MDS, AML, ALL, PMF or post-ET/PV MF in the last 3 - years prior to study inclusion).
* For healthy donors: previous or current hematological disease, previous or current other malignant disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hematological cancers: Adults (≥18 years) with MDS, AML, ALL, or primary/secondary myelofibrosis from whom blood and bone marrow samples will be collected during the disease course.
  Healthy donors: Adults (≥18 years) donating hematopoietic stem cells for allogeneic transplantation, providing peripheral blood or bone marrow samples as a source of healthy stem cells.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of metabolites | at primary diagnosis (month 0); after initial chemotherapy (month +0.5-2); before allo-HSCT (month +3-12); 1, 3, 6, 12 month after allo-HSCT (month 4-13, 6-15, 9-18, 15-24), and at relapse (if applicable, up to 5 years)
  the concentration of metabolites in malignant cells, immune cells, and extracellular fluid in each sample at the time point at which the sample is obtained. Metabolite and lipid concentrations will be measured by mass spectrometry.
Concentration of lipids | at primary diagnosis (month 0); after initial chemotherapy (month +0.5-2); before allo-HSCT (month +3-12); 1, 3, 6, 12 month after allo-HSCT (month 4-13, 6-15, 9-18, 15-24), and at relapse (if applicable, up to 5 years)
  the concentration of lipids in malignant cells, immune cells, and extracellular fluid in each sample at the time point at which the sample is obtained. Metabolite and lipid concentrations will be measured by mass spectrometry.
Expression profiling | at primary diagnosis (month 0); after initial chemotherapy (month +0.5-2); before allo-HSCT (month +3-12); 1, 3, 6, 12 month after allo-HSCT (month 4-13, 6-15, 9-18, 15-24), and at relapse (if applicable, up to 5 years)
  the expression of metabolite-related genes and proteins that will be measured by (single-cell) RNA-sequencing, quantitative polymerase chain reaction (PCR), proteomics, flow cytometry, western blotting, or another appropriate technique.
Metabolic function | at primary diagnosis (month 0); after initial chemotherapy (month +0.5-2); before allo-HSCT (month +3-12); 1, 3, 6, 12 month after allo-HSCT (month 4-13, 6-15, 9-18, 15-24), and at relapse (if applicable, up to 5 years)
  Metabolic function will be assessed by extracellular flux assays, flow cytometry, or another appropriate technique.

SECONDARY OUTCOMES:
Response to treatment(s) | during whole study, up to 5 years after allo-HSCT
Duration of the response | during whole study, up to 5 years after allo-HSCT
Progression-free survival | during whole study, up to 5 years after allo-HSCT
Overall survival | during whole study, up to 5 years after allo-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Petya Apostolova, Prof. Dr., Study Chair — University Hospital of Basel; Johannes Tossounidis, MD, Principal Investigator — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland